CLINICAL TRIAL: NCT00248989
Title: Effect of DHEA on Skin Aging - Placebo-Controlled and Randomized Phase III Study in Postmenopausal Women.
Brief Title: Effect of DHEA on Skin Aging in Postmenopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ERC-204
Record Dates: First submitted 2005-11-02; First posted 2005-11-04 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Skin Aging; Quality of Life
Keywords: Skin aging; Menopausal symptoms
MeSH Terms: interventions — Dehydroepiandrosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Experimental)
  Interventions: Drug: Placebos
- DHEA (Experimental)
  Interventions: Drug: Dehydroepiandrosterone

INTERVENTIONS:
Drug: Dehydroepiandrosterone — 3.0 ml of 0.3% DHEA cream applied on the skin twice daily.
  Arms: DHEA
Drug: Placebos — 3.0 ml of placebo cream applied on the skin twice daily.
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine the response of skin parameters related to skin aging to the local action of DHEA in postmenopausal women.

DETAILED DESCRIPTION:
Humans, along with the others primates, are unique among animal species in having adrenals that secrete large amounts of the inactive precursor steroids dehydroepiandrosterone(DHEA)and especially its sulfate DHEA-S. The marked reduction in the formation of DHEA-S by the adrenals during aging results in a dramatic fall in the formation of androgens and estrogens in peripheral target tissues, a situation that has been proposed to be associated with age-related diseases including skin atrophy, insulin resistance and obesity. Moreover, much attention has been given to the benefits of DHEA administered to postmenopausal women, especially on the bone, skin, vagina and well being after oral as well as percutaneous administration of the precursor steroid.

Therefore this study proposes to study the effect of 0.3% DHEA cream during a period of 12 months administered twice daily to postmenopausal women. During the study several biological and clinical parameters will be evaluated. In summary, these include blood steroid levels, distribution of hormonal receptors in the skin, sebaceous gland activity, skin hydration, skin wrinkles and finally skin genomic evaluation.

Subjects will be evaluated at specific time intervals for the above mentioned parameters as well as tolerability and adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy postmenopausal women who have taken hormonal replacement therapy for at least two years but not during the last 6 months prior to the study.
* Aged between 60 and 65.

Exclusion Criteria:

* Significant dermatologic, metabolic and endocrine disease.
* Diagnosis of cancer or history of hormone-dependant cancer.
* Over exposure to sun or tanning session during the previous two months.
* Narcotic addiction, alcoholism or smoking.

Ages: 60 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2004-11-01 (Actual); Primary Completion 2005-11-24 (Actual); Study Completion 2008-11-13 (Actual)

PRIMARY OUTCOMES:
Determination of local activity of DHEA for a 12 months period in parameters such as wrinkles, sebaceous gland activity, changes in skin morphology and other physical skin parameters.

SECONDARY OUTCOMES:
Evaluation of tolerance to local skin application of DHEA for a 12 months period and potential beneficial effects on quality of life including sexual life.

CONTACTS AND LOCATIONS:
Overall Officials: Leonello Cusan, MD, PhD, Principal Investigator — CHUL Research Center; Fernand Labrie, MD, PhD, Study Director — CHUL Research Center
Locations (1):
- Clinique des Traitements Hormonaux- CHUL Research Center, Sainte-Foy, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baulieu EE, Thomas G, Legrain S, Lahlou N, Roger M, Debuire B, Faucounau V, Girard L, Hervy MP, Latour F, Leaud MC, Mokrane A, Pitti-Ferrandi H, Trivalle C, de Lacharriere O, Nouveau S, Rakoto-Arison B, Souberbielle JC, Raison J, Le Bouc Y, Raynaud A, Girerd X, Forette F. Dehydroepiandrosterone (DHEA), DHEA sulfate, and aging: contribution of the DHEAge Study to a sociobiomedical issue. Proc Natl Acad Sci U S A. 2000 Apr 11;97(8):4279-84. doi: 10.1073/pnas.97.8.4279. PMID 10760294
- [Background] Bardon S, Vignon F, Chalbos D, Rochefort H. RU486, a progestin and glucocorticoid antagonist, inhibits the growth of breast cancer cells via the progesterone receptor. J Clin Endocrinol Metab. 1985 Apr;60(4):692-7. doi: 10.1210/jcem-60-4-692. PMID 3972969
- [Background] Belanger A, Candas B, Dupont A, Cusan L, Diamond P, Gomez JL, Labrie F. Changes in serum concentrations of conjugated and unconjugated steroids in 40- to 80-year-old men. J Clin Endocrinol Metab. 1994 Oct;79(4):1086-90. doi: 10.1210/jcem.79.4.7962278.
- [Background] Benz DJ, Haussler MR, Thomas MA, Speelman B, Komm BS. High-affinity androgen binding and androgenic regulation of alpha 1(I)-procollagen and transforming growth factor-beta steady state messenger ribonucleic acid levels in human osteoblast-like osteosarcoma cells. Endocrinology. 1991 Jun;128(6):2723-30. doi: 10.1210/endo-128-6-2723. PMID 2036957
- [Background] Burger HG, Hailes J, Menelaus M, Nelson J, Hudson B, Balazs N. The management of persistent menopausal symptoms with oestradiol-testosterone implants: clinical, lipid and hormonal results. Maturitas. 1984 Dec;6(4):351-8. doi: 10.1016/0378-5122(84)90008-2. PMID 6442755
- [Background] Casson PR, Andersen RN, Herrod HG, Stentz FB, Straughn AB, Abraham GE, Buster JE. Oral dehydroepiandrosterone in physiologic doses modulates immune function in postmenopausal women. Am J Obstet Gynecol. 1993 Dec;169(6):1536-9. doi: 10.1016/0002-9378(93)90431-h. PMID 8267058
- [Background] Chesnut CH 3rd, Ivey JL, Gruber HE, Matthews M, Nelp WB, Sisom K, Baylink DJ. Stanozolol in postmenopausal osteoporosis: therapeutic efficacy and possible mechanisms of action. Metabolism. 1983 Jun;32(6):571-80. doi: 10.1016/0026-0495(83)90027-6. PMID 6341772
- [Background] Colditz GA, Hankinson SE, Hunter DJ, Willett WC, Manson JE, Stampfer MJ, Hennekens C, Rosner B, Speizer FE. The use of estrogens and progestins and the risk of breast cancer in postmenopausal women. N Engl J Med. 1995 Jun 15;332(24):1589-93. doi: 10.1056/NEJM199506153322401. PMID 7753136
- [Background] Coleman DL, Leiter EH, Schwizer RW. Therapeutic effects of dehydroepiandrosterone (DHEA) in diabetic mice. Diabetes. 1982 Sep;31(9):830-3. doi: 10.2337/diab.31.9.830. PMID 6219024
- [Background] Davis SR, McCloud P, Strauss BJ, Burger H. Testosterone enhances estradiol's effects on postmenopausal bone density and sexuality. Maturitas. 1995 Apr;21(3):227-36. doi: 10.1016/0378-5122(94)00898-h. PMID 7616872
- [Background] DeFazio J, Meldrum DR, Winer JH, Judd HL. Direct action of androgen on hot flushes in the human male. Maturitas. 1984 Jul;6(1):3-8. doi: 10.1016/0378-5122(84)90060-4. PMID 6472125
- [Background] Diamond P, Cusan L, Gomez JL, Belanger A, Labrie F. Metabolic effects of 12-month percutaneous dehydroepiandrosterone replacement therapy in postmenopausal women. J Endocrinol. 1996 Sep;150 Suppl:S43-50. PMID 8943786
- [Background] El-Alfy M, Luu-The V, Huang XF, Berger L, Labrie F, Pelletier G. Localization of type 5 17beta-hydroxysteroid dehydrogenase, 3beta-hydroxysteroid dehydrogenase, and androgen receptor in the human prostate by in situ hybridization and immunocytochemistry. Endocrinology. 1999 Mar;140(3):1481-91. doi: 10.1210/endo.140.3.6585. PMID 10067877
- [Background] El-Alfy M, Pelletier G, Hermo LS, Labrie F. Unique features of the basal cells of human prostate epithelium. Microsc Res Tech. 2000 Dec 1;51(5):436-46. doi: 10.1002/1097-0029(20001201)51:53.0.CO;2-T. PMID 11074614
- [Background] Gordon GB, Shantz LM, Talalay P. Modulation of growth, differentiation and carcinogenesis by dehydroepiandrosterone. Adv Enzyme Regul. 1987;26:355-82. doi: 10.1016/0065-2571(87)90023-9. PMID 2960133
- [Background] Grodin JM, Siiteri PK, MacDonald PC. Source of estrogen production in postmenopausal women. J Clin Endocrinol Metab. 1973 Feb;36(2):207-14. doi: 10.1210/jcem-36-2-207. No abstract available. PMID 4688315
- [Background] Henderson E, Yang JY, Schwartz A. Dehydroepiandrosterone (DHEA) and synthetic DHEA analogs are modest inhibitors of HIV-1 IIIB replication. AIDS Res Hum Retroviruses. 1992 May;8(5):625-31. doi: 10.1089/aid.1992.8.625. PMID 1381206
- [Background] HENNEMAN PH, WALLACH S. A review of the prolonged use of estrogens and androgens in postmenopausal and senile osteoporosis. AMA Arch Intern Med. 1957 Nov;100(5):715-23. doi: 10.1001/archinte.1957.00260110031005. No abstract available. PMID 13468816
- [Background] Johnston CC Jr, Epstein S. Clinical, biochemical, radiographic, epidemiologic, and economic features of osteoporosis. Orthop Clin North Am. 1981 Jul;12(3):559-69. PMID 7290587
- [Background] Johnston CC Jr, Hui SL, Witt RM, Appledorn R, Baker RS, Longcope C. Early menopausal changes in bone mass and sex steroids. J Clin Endocrinol Metab. 1985 Nov;61(5):905-11. doi: 10.1210/jcem-61-5-905. PMID 3930555
- [Background] Kapur SP, Reddi AH. Influence of testosterone and dihydrotestosterone on bone-matrix induced endochondral bone formation. Calcif Tissue Int. 1989 Feb;44(2):108-13. doi: 10.1007/BF02556469. PMID 2492887
- [Background] Labrie C, Belanger A, Labrie F. Androgenic activity of dehydroepiandrosterone and androstenedione in the rat ventral prostate. Endocrinology. 1988 Sep;123(3):1412-7. doi: 10.1210/endo-123-3-1412. PMID 2969802
- [Background] Labrie F. Intracrinology. Mol Cell Endocrinol. 1991 Jul;78(3):C113-8. doi: 10.1016/0303-7207(91)90116-a. PMID 1838082
- [Background] Labrie F, Belanger A, Cusan L, Candas B. Physiological changes in dehydroepiandrosterone are not reflected by serum levels of active androgens and estrogens but of their metabolites: intracrinology. J Clin Endocrinol Metab. 1997 Aug;82(8):2403-9. doi: 10.1210/jcem.82.8.4161. PMID 9253308
- [Background] Labrie F, Belanger A, Cusan L, Gomez JL, Candas B. Marked decline in serum concentrations of adrenal C19 sex steroid precursors and conjugated androgen metabolites during aging. J Clin Endocrinol Metab. 1997 Aug;82(8):2396-402. doi: 10.1210/jcem.82.8.4160. PMID 9253307
- [Background] Labrie F, Belanger A, Simard J, Van Luu-The, Labrie C. DHEA and peripheral androgen and estrogen formation: intracinology. Ann N Y Acad Sci. 1995 Dec 29;774:16-28. doi: 10.1111/j.1749-6632.1995.tb17369.x. No abstract available. PMID 8597456
- [Background] Labrie F, Diamond P, Cusan L, Gomez JL, Belanger A, Candas B. Effect of 12-month dehydroepiandrosterone replacement therapy on bone, vagina, and endometrium in postmenopausal women. J Clin Endocrinol Metab. 1997 Oct;82(10):3498-505. doi: 10.1210/jcem.82.10.4306. PMID 9329392
- [Background] Labrie F, Luu-The V, Labrie C, Belanger A, Simard J, Lin SX, Pelletier G. Endocrine and intracrine sources of androgens in women: inhibition of breast cancer and other roles of androgens and their precursor dehydroepiandrosterone. Endocr Rev. 2003 Apr;24(2):152-82. doi: 10.1210/er.2001-0031. PMID 12700178
- [Background] Labrie F, Luu-The V, Lin SX, Labrie C, Simard J, Breton R, Belanger A. The key role of 17 beta-hydroxysteroid dehydrogenases in sex steroid biology. Steroids. 1997 Jan;62(1):148-58. doi: 10.1016/s0039-128x(96)00174-2. PMID 9029730
- [Background] Labrie F, Luu-The V, Lin SX, Simard J, Labrie C. Role of 17 beta-hydroxysteroid dehydrogenases in sex steroid formation in peripheral intracrine tissues. Trends Endocrinol Metab. 2000 Dec;11(10):421-7. doi: 10.1016/s1043-2760(00)00342-8. PMID 11091120
- [Background] Labrie F, Simard J, Luu-The V, Bélanger A, Pelletier G, Morel Y, Mebarki F, Sanchez R, Durocher F, Turgeon C, Labrie Y, Rhéaume E, Labrie C, Lachance Y. The 3b-hydroxysteroid dehydrogenase/isomerase gene family: lessons from type II 3b-HSD congenital deficiency. In: Signal Transduction in Testicular Cells. Ernst Schering Research Foundation Workshop. Hansson V, Levy FO, Taskén K (eds), Berlin, Heidelberg, New York, Springer-Verlag, Vol. Suppl. 2: pp. 185-218, 1996.
- [Background] Leiblum S, Bachmann G, Kemmann E, Colburn D, Swartzman L. Vaginal atrophy in the postmenopausal woman. The importance of sexual activity and hormones. JAMA. 1983 Apr 22-29;249(16):2195-8. PMID 6834616
- [Background] Li S, Yan X, Belanger A, Labrie F. Prevention by dehydroepiandrosterone of the development of mammary carcinoma induced by 7,12-dimethylbenz(a)anthracene (DMBA) in the rat. Breast Cancer Res Treat. 1994 Feb;29(2):203-17. doi: 10.1007/BF00665681. PMID 8012037
- [Background] MacEwen EG, Kurzman ID. Obesity in the dog: role of the adrenal steroid dehydroepiandrosterone (DHEA). J Nutr. 1991 Nov;121(11 Suppl):S51-5. doi: 10.1093/jn/121.suppl_11.S51. PMID 1834816
- [Background] Mazess RB. On aging bone loss. Clin Orthop Relat Res. 1982 May;(165):239-52. PMID 7075066
- [Background] MIGEON CJ, KELLER AR, LAWRENCE B, SHEPARD TH 2nd. Dehydroepiandrosterone and androsterone levels in human plasma: effect of age and sex; day-to-day and diurnal variations. J Clin Endocrinol Metab. 1957 Sep;17(9):1051-62. doi: 10.1210/jcem-17-9-1051. No abstract available. PMID 13463066
- [Background] Morales AJ, Nolan JJ, Nelson JC, Yen SS. Effects of replacement dose of dehydroepiandrosterone in men and women of advancing age. J Clin Endocrinol Metab. 1994 Jun;78(6):1360-7. doi: 10.1210/jcem.78.6.7515387.
- [Background] Need AG, Horowitz M, Bridges A, Morris HA, Nordin BE. Effects of nandrolone decanoate and antiresorptive therapy on vertebral density in osteoporotic postmenopausal women. Arch Intern Med. 1989 Jan;149(1):57-60. PMID 2912415
- [Background] Nestler JE, Barlascini CO, Clore JN, Blackard WG. Dehydroepiandrosterone reduces serum low density lipoprotein levels and body fat but does not alter insulin sensitivity in normal men. J Clin Endocrinol Metab. 1988 Jan;66(1):57-61. doi: 10.1210/jcem-66-1-57. PMID 2961787
- [Background] Notelovitz M, Watts N, Timmons C, Addison A, Wiita B, Downey L. Effects of estrogen plus low dose androgen vs estrogen alone on menopausal symptoms in oophorectomized/hysterectomized. North Am. Menopause Soc., Montreal 1991, 101.
- [Background] Orentreich N, Brind JL, Rizer RL, Vogelman JH. Age changes and sex differences in serum dehydroepiandrosterone sulfate concentrations throughout adulthood. J Clin Endocrinol Metab. 1984 Sep;59(3):551-5. doi: 10.1210/jcem-59-3-551. PMID 6235241
- [Background] Pye JK, Mansel RE, Hughes LE. Clinical experience of drug treatments for mastalgia. Lancet. 1985 Aug 17;2(8451):373-7. doi: 10.1016/s0140-6736(85)92506-1. PMID 2862523
- [Background] Rasmussen KR, Arrowood MJ, Healey MC. Effectiveness of dehydroepiandrosterone in reduction of cryptosporidial activity in immunosuppressed rats. Antimicrob Agents Chemother. 1992 Jan;36(1):220-2. doi: 10.1128/AAC.36.1.220. PMID 1534212
- [Background] Riggs BL, Wahner HW, Dunn WL, Mazess RB, Offord KP, Melton LJ 3rd. Differential changes in bone mineral density of the appendicular and axial skeleton with aging: relationship to spinal osteoporosis. J Clin Invest. 1981 Feb;67(2):328-35. doi: 10.1172/JCI110039. PMID 7462421
- [Background] Savvas M, Studd JW, Fogelman I, Dooley M, Montgomery J, Murby B. Skeletal effects of oral oestrogen compared with subcutaneous oestrogen and testosterone in postmenopausal women. BMJ. 1988 Jul 30;297(6644):331-3. doi: 10.1136/bmj.297.6644.331. PMID 3137998
- [Background] Schriock ED, Buffington CK, Hubert GD, Kurtz BR, Kitabchi AE, Buster JE, Givens JR. Divergent correlations of circulating dehydroepiandrosterone sulfate and testosterone with insulin levels and insulin receptor binding. J Clin Endocrinol Metab. 1988 Jun;66(6):1329-31. doi: 10.1210/jcem-66-6-1329. PMID 2967305
- [Background] Schwartz AG, Pashko L, Whitcomb JM. Inhibition of tumor development by dehydroepiandrosterone and related steroids. Toxicol Pathol. 1986;14(3):357-62. doi: 10.1177/019262338601400312. PMID 3024302
- [Background] Sherwin BB. Affective changes with estrogen and androgen replacement therapy in surgically menopausal women. J Affect Disord. 1988 Mar-Apr;14(2):177-87. doi: 10.1016/0165-0327(88)90061-4. PMID 2966832
- [Background] Sherwin BB, Gelfand MM. Effects of parenteral administration of estrogen and androgen on plasma hormone levels and hot flushes in the surgical menopause. Am J Obstet Gynecol. 1984 Mar 1;148(5):552-7. doi: 10.1016/0002-9378(84)90746-4. PMID 6367474
- [Background] Sherwin BB, Gelfand MM. Differential symptom response to parenteral estrogen and/or androgen administration in the surgical menopause. Am J Obstet Gynecol. 1985 Jan 15;151(2):153-60. doi: 10.1016/0002-9378(85)90001-8. PMID 3881960
- [Background] Sherwin BB, Gelfand MM. The role of androgen in the maintenance of sexual functioning in oophorectomized women. Psychosom Med. 1987 Jul-Aug;49(4):397-409. doi: 10.1097/00006842-198707000-00009. PMID 3615768
- [Background] Sourla A, Richard V, Labrie F, Labrie C. Exclusive androgenic effect of dehydroepiandrosterone in sebaceous glands of rat skin. J Endocrinol. 2000 Aug;166(2):455-62. doi: 10.1677/joe.0.1660455. PMID 10927635
- [Background] Steinberg KK, Freni-Titulaer LW, DePuey EG, Miller DT, Sgoutas DS, Coralli CH, Phillips DL, Rogers TN, Clark RV. Sex steroids and bone density in premenopausal and perimenopausal women. J Clin Endocrinol Metab. 1989 Sep;69(3):533-9. doi: 10.1210/jcem-69-3-533. PMID 2527242
- [Background] Studd J W, Collins W P, Chakravarti S, Newton J R, Oram D, Parsons A. Estradiol and testosterone implants in treatment of psochosexual problems in postmenopausal women. Br. J. Obstet. Gynecol. 84: 314-315, 1987.
- [Background] Suzuki T, Suzuki N, Daynes RA, Engleman EG. Dehydroepiandrosterone enhances IL2 production and cytotoxic effector function of human T cells. Clin Immunol Immunopathol. 1991 Nov;61(2 Pt 1):202-11. doi: 10.1016/s0090-1229(05)80024-8. PMID 1833106
- [Background] Tchernof A, Despres JP, Belanger A, Dupont A, Prud'homme D, Moorjani S, Lupien PJ, Labrie F. Reduced testosterone and adrenal C19 steroid levels in obese men. Metabolism. 1995 Apr;44(4):513-9. doi: 10.1016/0026-0495(95)90060-8. PMID 7723675
- [Background] Vermeulen A, Deslypere JP, Schelfhout W, Verdonck L, Rubens R. Adrenocortical function in old age: response to acute adrenocorticotropin stimulation. J Clin Endocrinol Metab. 1982 Jan;54(1):187-91. doi: 10.1210/jcem-54-1-187. PMID 6274897
- [Background] Vermeulen A, Verdonck L. Radioimmunoassay of 17beta-hydroxy-5alpha-androstan-3-one, 4-androstene-3,17-dione, dehydroepiandrosterone, 17-hydroxyprogesterone and progesterone and its application to the human male plasma. J Steroid Biochem. 1976 Jan;7(1):1-10. doi: 10.1016/0022-4731(76)90156-4. No abstract available. PMID 178963
- [Background] Zumoff B, Strain GW, Miller LK, Rosner W. Twenty-four-hour mean plasma testosterone concentration declines with age in normal premenopausal women. J Clin Endocrinol Metab. 1995 Apr;80(4):1429-30. doi: 10.1210/jcem.80.4.7714119.
- [Result] Labrie F, Cusan L, Gomez JL, Martel C, Berube R, Belanger P, Chaussade V, Deloche C, Leclaire J. Changes in serum DHEA and eleven of its metabolites during 12-month percutaneous administration of DHEA. J Steroid Biochem Mol Biol. 2008 May;110(1-2):1-9. doi: 10.1016/j.jsbmb.2008.02.003. Epub 2008 Feb 14. PMID 18359622